CLINICAL TRIAL: NCT06804252
Title: Incidence of Fragility Fractures and Osteoporosis Screening in Chronic Stroke Patients: a Prospective Observational Study
Brief Title: Incidence of Fragility Fractures and Osteoporosis Screening in Chronic Stroke Patients
Status: Active, not recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Other Study IDs: MFR022025
Record Dates: First submitted 2025-01-18; First posted 2025-02-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Chronic Stroke; Osteoporosis; Fragility Fractures
Keywords: chronic stroke; osteoporis; fragility fractures; Hip fractures; Stroke risk factors; Bone density (DEXA); bone; Bone mineral density; Bone metabolism; Bone health; Bone health intervention; Post-stroke; Bone density screening
MeSH Terms: conditions — Osteoporosis; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Stroke Patients Aged 65 and Above: This group consists of patients aged 65 years and older who have experienced a chronic stroke. These patients are assessed for the incidence of osteoporosis and fragility fractures, and are evaluated for bone metabolism management following the cerebrovascular event. The study aims to determine the prevalence of osteoporosis and fractures, as well as the effectiveness of screening for bone metabolism disorders in this specific population.

SUMMARY:
Stroke is a known risk factor for the development of osteoporosis, leading to an increased risk of falls and fractures. Several international studies have associated stroke with hip fractures, showing an odds ratio ranging between 1.5 and 4. The literature frequently indicates a lack of management for bone metabolism in patients following cerebrovascular events. This study aims to evaluate the incidence of osteoporosis and fragility fractures in patients with chronic stroke. A secondary aim is to assess whether patients have been adequately screened for bone metabolism following a cerebrovascular event. This study is designed as a prospective observational study. Patients aged over 65 years with chronic stroke are assessed at the U.O.C. of "Functional Recovery and Rehabilitation" at A.O.U.P. "P. Giaccone," Palermo. During the assessment, clinical and demographic data are collected, including details of the cerebrovascular event (location, hemorrhagic/ischemic, date), pre-event and post-event disability/autonomy (Rankin scale), presence of fractures (location and date) in the patient's medical history (pre and post-event), femoral and lumbar DEXA for osteoporosis evaluation, and DeFRA for assessing the 10-year risk of fragility fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older
* Diagnosed with chronic stroke
* Able to provide informed consent
* Willing to participate in follow-up assessments
* Stable medical condition that allows participation in the study

Exclusion Criteria:

* Patients with acute stroke
* Severe cognitive impairment that prevents informed consent
* Other major illnesses affecting bone metabolism (e.g., severe renal disease)
* Patients already undergoing treatment for osteoporosis
* Patients with conditions that contraindicate DEXA scan

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Study Population: Participants will be selected from patients aged 65 and older who have experienced a chronic stroke and are receiving treatment at the Neurology and Rehabilitation Departments of hospitals in Palermo, Italy. The population includes both male and female patients who meet the inclusion criteria and are willing to provide informed consent. The study aims to evaluate the incidence of osteoporosis and fragility fractures in this specific population and to assess their bone metabolism management post-cerebrovascular event.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluating the Incidence of Osteoporosis and Fragility Fractures in Chronic Stroke Patients | From enrollment to the end of treatment at 6 months
  The primary objective of this study is to evaluate the incidence of osteoporosis and fragility fractures in patients with chronic stroke.

SECONDARY OUTCOMES:
Proper screening for bone metabolism in patients after cerebrovascular event | From enrollment to the end of treatment at 6 months
  Number of patients who were properly screened for bone metabolism after the cerebrovascular event.

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U.P. P. Giaccone, Palermo, Italia 90127, Palermo, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code